CLINICAL TRIAL: NCT02227225
Title: Factors Affecting the Incidence of Postoperative Delirium in Frail Elderly Undergoing Non-cardiac Surgery: An Observational Study
Brief Title: Factors Affecting the Incidence of Postoperative Delirium in Frail Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Shariq Ali Khan, Consultant, Singapore General Hospital
Other Study IDs: C2014/748
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Postoperative Delirium
Keywords: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postoperative Delirium

SUMMARY:
Postoperative delirium has been found to be associated with increased risk of future neurocognitive decline and mortality especially in elderly patients. Similarly, Frailty has been found to be associated with an increased risk of postoperative complication including delirium in the elderly.The purpose of this study is determine the factors affecting the incidence of postoperative delirium in frail elderly undergoing non-cardiac surgery in the Singapore population.

ELIGIBILITY:
Inclusion Criteria:

* Elderly (> 65 years) frail patients undergoing non cardiac surgery under anaesthesia lasting for >60 minutes
* Patient willing and able to complete the requirements of this study.

Exclusion Criteria:

* disabling neuropsychiatric or neurological disorders(including severe dementia, Alzheimer's disease, schizophrenia, severe depression)
* patients suffering from delirium at selection;
* patients who cannot complete the preoperative mental tests (CAM and/or Mini-Mental State Examination (MMSE)) of this clinical trial;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Postoperative inpatients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
postoperative delirium | upto 3 postoperative days
  Confusion assessment method (CAM) will be used to asses delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore